CLINICAL TRIAL: NCT01572948
Title: A Placebo-controlled Trial of Roflumilast (Daliresp) on Markers of Inflammation in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Placebo-controlled Trial of Daliresp on Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, J Edwin Blalock, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAL-MD-01
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Results first posted 2015-07-31 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo (Forest Laboratories, Inc) is manufactured as an odorless and otherwise equivalent tablet to the roflumilast tablet, but contains no active ingredient.
  Interventions: Drug: placebo
- Daliresp (Active Comparator): The study drug (roflumilast, Daliresp™, Forest Laboratories, Inc.) is a targeted inhibitor of phosphodiesterase 4 and is given once daily via oral route. There is proven anti-inflammatory and anti-oxidant potential in both animal and human models
  Interventions: Drug: roflumilast

INTERVENTIONS:
Drug: roflumilast — The study drug (roflumilast, Daliresp™, Forest Laboratories, Inc.) is a targeted inhibitor of phosphodiesterase 4 and is given once daily via oral route. There is proven anti-inflammatory and anti-oxidant potential in both animal and human models
  Other Names: Daliresp
  Arms: Daliresp
Drug: placebo — The placebo (Forest Laboratories, Inc) is manufactured as an odorless and otherwise equivalent tablet to the roflumilast tablet, but contains no active ingredient
  Arms: Placebo

SUMMARY:
The purpose of the study is to propose that roflumilast is associated with meaningful reductions in biomarkers of pulmonary inflammation and sputum neutrophilia, including confirmation of previously described results, and correlate these findings with improvement in pulmonary function, sputum scores, and quality of life in stable moderate to severe COPD. The investigators aim to demonstrate this regardless of concomitant medication use, including inhaled corticosteroids. Additionally, the investigators hope to provide a mechanistic pathway by which these effects occur.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, > 40 years of age
2. Clinical diagnosis of moderate to severe COPD as defined by the GOLD criteria:

   Post-bronchodilator FEV1/FVC < 70% Post-bronchodilator FEV1 < 70% predicted
3. Cigarette consumption of 10 pack-years or more. Patients may be active smokers.
4. The presence of chronic cough and sputum production
5. Willingness to make return visits and telephone availability for the study duration

Exclusion Criteria:

1. A diagnosis of asthma as established by the study investigator on the basis of the recent American Thoracic Society/European Respiratory Society guidelines
2. Clinically significant bronchiectasis
3. Oxygen use >12 hours/day
4. Known sensitivity to roflumilast
5. Use of other methylxanthines within 1 month (theophylline)
6. Changes to current maintenance COPD therapy within one month
7. Pregnancy
8. An acute illness requiring antibiotics and/or corticosteroids within the month prior to enrolment.
9. Immunosuppression

   1. HIV
   2. Solid organ transplant
   3. Active malignancy
   4. Systemic corticosteroid use ≥ prednisone 20mg / day
   5. Other immunosuppressants
10. Terminal illness defined as anticipated survival <12 months
11. Severe comorbidities including uncontrolled angina, congestive heart failure, end-stage renal disease, liver failure, or other conditions that would preclude the patient from safely completing the required tests or the study.

    -

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Blalock, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Lung Health Center, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Wells JM, Jackson PL, Viera L, Bhatt SP, Gautney J, Handley G, King RW, Xu X, Gaggar A, Bailey WC, Dransfield MT, Blalock JE. A Randomized, Placebo-controlled Trial of Roflumilast. Effect on Proline-Glycine-Proline and Neutrophilic Inflammation in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2015 Oct 15;192(8):934-42. doi: 10.1164/rccm.201503-0543OC. PMID 26151090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a single center.
Groups:
- Roflumilast: group randomized to 30 day supply of white tablet 500microgram
- Placebo: 500microgram white tablet
Period: Overall Study
Arm/Group | Roflumilast | Placebo
Started | 11 | 16
Completed | 10 | 15
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — unable to contact | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Roflumilast | Total
Number analyzed (Participants) | 16 | 11 | 27
Age, Continuous [Mean (Full Range); unit: years] | 61 [53 to 69] | 62 [55 to 69] | 61 [53 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 10 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 12 | 7 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 11 | 27

OUTCOME MEASURES:

1. Primary Outcome: Induced Sputum Proline-glycine-proline (PGP) Levels at Baseline
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Roflumilast
Number analyzed (Participants) | 16 | 11
ng/ml | 0.74 (0.25) | 0.64 (0.21)

2. Secondary Outcome: Induced Sputum Neutrophil Count
Time Frame: 1 month
Measure: Mean (Standard Error); unit: percentage of sputum neutrophils
Arm/Group | Placebo | Daliresp
Number analyzed (Participants) | 16 | 11
percentage of sputum neutrophils | 83 (.24) | 80 (.24)

3. Primary Outcome: Mean Induced Sputum Proline-glycine-proline (PGP) Levels at 1 Month After Randomization.
Time Frame: 1 month after baseline
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 11 | 16
ng/ml | .33 (.12) | .66 (.18)

4. Primary Outcome: Mean Induced Sputum Proline-glycine-proline (PGP) Levels at 3 Months After Randomization
Time Frame: 3 months after baseline
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Roflumilast
Number analyzed (Participants) | 16 | 11
ng/ml | 0.70 (0.18) | 0.30 (0.11)

5. Secondary Outcome: Induced Sputum Neutrophil Count
Time Frame: baseline
Measure: Mean (Standard Error); unit: percentage of sputum neutrophils
Arm/Group | Placebo | Roflumilast
Number analyzed (Participants) | 16 | 11
percentage of sputum neutrophils | 89 (.25) | 83 (.23)

6. Secondary Outcome: Induced Sputum Neutrophil Count
Time Frame: 3 months after baseline
Measure: Mean (Standard Error); unit: percentage of sputum neutrophils
Arm/Group | Placebo | Roflumilast
Number analyzed (Participants) | 16 | 11
percentage of sputum neutrophils | 86 (.24) | 58 (.18)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | Roflumilast
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/11
Other Adverse Events (participants affected / at risk) | 4/16 | 5/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Roflumilast (N=11)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
weight loss of 10lbs (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pleurisy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
insomnia (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
small sample size and limited follow-up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No